CLINICAL TRIAL: NCT03816059
Title: Respiratory Virus Infections in Acutely Hospitalized Adult Patients With Pulmonary and Extrapulmonary Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: 20190104
Record Dates: First submitted 2019-01-15; First posted 2019-01-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Virus Infection; Stroke; Lung Disease; Acute Coronary Syndrome
Keywords: Respiratory virus infection; Extrapulmonary complications; Myocardial infarction; Asthma; Bronchiectasis; Chronic obstructive pulmonary disease; Cerebrovascular disease
MeSH Terms: conditions — Stroke; Lung Diseases; Acute Coronary Syndrome; Myocardial Infarction; Asthma; Bronchiectasis; Pulmonary Disease, Chronic Obstructive; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva specimens will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hospitalized - ACS: Hospitalized patients with acute coronary syndrome
  Interventions: Diagnostic Test: Respiratory virus testing
- Hospitalized - stroke: Hospitalized patients with stroke
  Interventions: Diagnostic Test: Respiratory virus testing
- Hospitalized - chronic lung disease: Hospitalized patients with exacerbation of chronic lung disease
  Interventions: Diagnostic Test: Respiratory virus testing
- Outpatient: Outpatients
  Interventions: Diagnostic Test: Respiratory virus testing

INTERVENTIONS:
Diagnostic Test: Respiratory virus testing — All patients will be tested for respiratory viruses

SUMMARY:
Respiratory virus infections are one of the major causes of hospitalizations, and outbreaks of respiratory virus infection have led to severe economic loss. In addition to pulmonary complications, respiratory viruses can also lead to non-pulmonary complications.

However, many previous studies on the complications of respiratory viruses are retrospective in nature, and therefore many patients with respiratory virus infection may not be tested. Furthermore, these studies did not take into account that respiratory viruses can be found in some asymptomatic individuals. The aim of this study is to capture the burden of respiratory viruses in patients with acute pulmonary and extrapulmonary complications. We will recruit patients admitted to our hospital with acute coronary syndrome, stroke and exacerbation of underlying lung diseases. We will collect saliva from these patients and test for respiratory viruses. As controls, we will recruit asymptomatic patients at the out-patient clinic for follow up of chronic heart, lung or neurological diseases.

We anticipate that this study will greatly enhance our understanding of the epidemiology of respiratory viruses in acutely hospitalized patients. Our findings will be important for clinicians, public health practitioners and scientists.

DETAILED DESCRIPTION:
Respiratory viruses cause severe infections, and contribute to a substantial number of hospitalizations, admission to intensive care units and deaths. Many hospitalizations due to respiratory virus infection are related to pneumonia or exacerbation of chronic lung disease. In addition, many hospitalizations are related to extrapulmonary complications, such as acute coronary syndrome or stroke.

Previous studies have reported the incidence of respiratory viruses among patients with pulmonary complications, or the association of respiratory viruses with acute coronary syndrome or stroke. However, there are several problems associated with these studies. First, many of these studies are retrospective in nature, and therefore testing was only performed in selected patients with respiratory symptoms. Hence, many patients without respiratory symptoms were not recruited. Second, respiratory virus can be detected in some asymptomatic individuals. Therefore, the presence of respiratory virus may be an incidental finding rather than the cause of the complication. Third, many studies only focus on a few respiratory viruses, especially on influenza virus.

This study aims to address these issues. The investigators propose to conduct a prospective cohort study. The investigators will recruit hospitalized adult patients with exacerbation of underlying lung disease, acute coronary syndrome or stroke. As controls, the investigators will recruit outpatients follow-up for chronic heart disease, chronic lung disease or neurological conditions. The investigators will collect saliva from study participants and perform respiratory virus testing using a multiplex PCR panel. Previous studies have shown that there is a high concordance between results from respiratory virus testing on saliva and nasopharyngeal specimens. The investigators will also use a standardized questionnaire to collect information regarding symptoms.

This study will provide accurate data on the epidemiology of respiratory viruses in pulmonary and extrapulmonary complications.These data are important for clinicians, public health practitioners and scientists.

ELIGIBILITY:
Inclusion Criteria: (For hospitalized patients)

1. Admitted to the acute medical ward of Queen Mary Hospital via the accident and emergency department
2. Aged 18 years or above
3. Hospitalized for less than 24 hours at the time of recruitment
4. Presented with exacerbation of underlying lung disease, acute coronary syndrome or stroke
5. Competent and agree to provide written informed consent

Exclusion Criteria: (For hospitalized patients)

1. Admitted to any hospitals in the past 14 days
2. Respiratory virus testing performed in the past 14 days
3. Antiviral against respiratory virus given within the past 14 days
4. Not sufficient saliva

Inclusion Criteria: (For out-patients)

1. Aged 18 years or above
2. Follow-up at out-patient clinic or at the physiotherapy department of Queen Mary Hospital
3. Competent and agree to provide written informed consent

Exclusion criteria: (For out-patients)

1. Admitted to any hospitals in the past 14 days
2. Respiratory virus testing performed in the past 14 days
3. Antiviral against respiratory virus given within the past 14 days
4. Onset of new respiratory or non-respiratory symptoms within the past 14 days
5. Not sufficient saliva

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Hospitalized patients with acute coronary syndrome, stroke or exacerbation of underlying lung disease
  2. Outpatients follow-up for chronic conditions
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory viruses | 2 days
  Incidence of respiratory viruses

SECONDARY OUTCOMES:
Length of hospital stay | 1 month
  Length of hospital stay
Length of stay in general medical ward | 1 month
  Length of stay in general medical ward
Length of stay in high dependency unit | 1 month
  Length of stay in high dependency unit
Length of stay in intensive care unit | 1 month
  Length of stay in intensive care unit
Proportion of patients requiring oxygen supplementation | 1 month
  Proportion of patients requiring oxygen supplementation
Proportion of patients requiring positive pressure ventilation | 1 month
  Proportion of patients requiring positive pressure ventilation
Proportion of patients requiring intubation | 1 month
  Proportion of patients requiring intubation
Proportion of patients admitted to intensive care unit | 1 month
  Proportion of patients admitted to intensive care unit
Proportion of patients admitted to coronary care unit | 1 month
  Proportion of patients admitted to coronary care unit
Proportion of patients admitted to high dependency unit | 1 month
  Proportion of patients admitted to high dependency unit
Proportion of patients who die during hospitalization | 1 month
  Proportion of patients who die during hospitalization
White blood cell on admission | 1 day
  White blood cell count in blood (x 10^9 cells/L)
Platelet count upon admission | 1 day
  Platelet count in blood (x 10^9 cells/L) upon admission
Alanine aminotransferase upon admission | 1 day
  The level of alanine aminotransferase in blood (U/L)
Creatinine on admission | 1 day
  The level of creatinine in blood (umol/L) upon
Blood culture result | 3 days
  The result of blood culture
Sputum culture result | 3 days
  The result of sputum culture
Proportion of patients with pneumonia | 1 month
  Proportion of patients with pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sellers SA, Hagan RS, Hayden FG, Fischer WA 2nd. The hidden burden of influenza: A review of the extra-pulmonary complications of influenza infection. Influenza Other Respir Viruses. 2017 Sep;11(5):372-393. doi: 10.1111/irv.12470. PMID 28745014
- [Result] To KK, Lau SK, Chan KH, Mok KY, Luk HK, Yip CC, Ma YK, Sinn LH, Lam SH, Ngai CW, Hung IF, Chan KH, Yuen KY. Pulmonary and extrapulmonary complications of human rhinovirus infection in critically ill patients. J Clin Virol. 2016 Apr;77:85-91. doi: 10.1016/j.jcv.2016.02.014. Epub 2016 Feb 20. PMID 26921740
- [Result] Warren-Gash C, Blackburn R, Whitaker H, McMenamin J, Hayward AC. Laboratory-confirmed respiratory infections as triggers for acute myocardial infarction and stroke: a self-controlled case series analysis of national linked datasets from Scotland. Eur Respir J. 2018 Mar 29;51(3):1701794. doi: 10.1183/13993003.01794-2017. Print 2018 Mar. PMID 29563170
- [Result] To KK, Lu L, Yip CC, Poon RW, Fung AM, Cheng A, Lui DH, Ho DT, Hung IF, Chan KH, Yuen KY. Additional molecular testing of saliva specimens improves the detection of respiratory viruses. Emerg Microbes Infect. 2017 Jun 7;6(6):e49. doi: 10.1038/emi.2017.35. PMID 28588283
- [Result] To KKW, Yip CCY, Lai CYW, Wong CKH, Ho DTY, Pang PKP, Ng ACK, Leung KH, Poon RWS, Chan KH, Cheng VCC, Hung IFN, Yuen KY. Saliva as a diagnostic specimen for testing respiratory virus by a point-of-care molecular assay: a diagnostic validity study. Clin Microbiol Infect. 2019 Mar;25(3):372-378. doi: 10.1016/j.cmi.2018.06.009. Epub 2018 Jun 12. PMID 29906597

DOCUMENTS (2):
  • Informed Consent Form (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03816059/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03816059/Prot_SAP_001.pdf